CLINICAL TRIAL: NCT00151515
Title: A Double-Blind, Randomized, Placebo-Controlled Trial of the Efficacy and Safety of 5 Percent Minoxidil Foam in the Treatment of Androgenetic Alopecia in Males
Brief Title: A Study to Evaluate the Effectiveness and Safety of 5 Percent Minoxidil Foam in the Treatment of Male Pattern Hair Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6221001
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Androgenetic Alopecia
Keywords: Alopecia, Balding
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Topical 5% minoxidil foam formulation used twice daily
  Interventions: Drug: minoxidil

INTERVENTIONS:
Drug: minoxidil — Topical 5% minoxidil foam, BID, for sixteen weeks
  Other Names: Formula # P902942A00 vs Placebo foam (Formula # P902943A00)

SUMMARY:
The primary purpose of the study is to evaluate the efficacy of a topical 5% minoxidil formulation in males for the treatment of pattern hair loss. The secondary purpose is to evaluate the safety of a topical 5% minoxidil formulation in males when used twice daily for the treatment of pattern hair loss and to obtain the safety data on the investigational product when used twice daily for up to one year.

DETAILED DESCRIPTION:
Male subjects with androgenetic alopecia were enrolled in this fourteen-center trial. Subjects were randomized to use either 5% minoxidil or placebo foam twice daily for 16 weeks. A total of 143 subjects continued use of the 5% minoxidil foam for 8 to 12 months in an open-label phase to obtain safety data on 5% minoxidil topical foam when used twice daily for up to one year.

The 5% minoxidil foam was shown to be effective in the treatment of male androgenetic alopecia in a 16 week trial. It was statistically significantly superior to placebo foam in the primary efficacy measure of mean change in the non-vellus hair count in the target region between Baseline and Week 16, and the subject rating assessed an overall improvement from Baseline.

The efficacy of 5% minoxidil compared to placebo was confirmed by the secondary efficacy endpoints of scores from the expert panel review of hair regrowth when comparing photographs obtained at Baseline with photographs obtained at Week 16, as well as the percent change from Baseline in non-vellus hair counts within a pre-specified area of clipped hair.

The 5% minoxidil foam formulation was well tolerated, the incidence of adverse events was similar between groups, and no safety concerns were raised based on clinical laboratory test results, vital signs or scalp irritation scores.

ELIGIBILITY:
Inclusion Criteria:

* presence of androgenetic alopecia with vertex pattern IIIv, IV, or V on the Norwood Hamilton Scale
* Male sex, age 15 to 49, good health
* Willingness to have a dot tattoo placed in the target area of the scalp during the study
* Willingness to maintain normal shampooing habits and products during the study
* Willingness to maintain the same hair style, approximate length, and hair color throughout the study

Exclusion Criteria:

* Known sensitivity to the investigational product

Ages: 15 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 352 (Actual)
Dates: Start 2003-10; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Mean change in non-vellus hair count in the target region as determined by validated computer-assisted dot-mapping technique and subject ratings | Baseline to 16 Weeks

SECONDARY OUTCOMES:
Visual assessment of local dermatitis | Each visit, Baseline through Week 16
Vital Signs | Each visit, Baseline through Week 16
Secondary efficacy evaluated by expert panel review of hair regrowth when comparing global photographs | Baseline vs Week 16
Percent change from baseline in non-vellus hair counts within a specified area of clipped hair | Baseline vs Week 16
Adverse Events | Each visit, Baseline through Week 16
Laboratory Tests (hematology, chemistries, and urinalysis) | at Baseline, Week 8, and Week 16 and Final Visit
Clinical safety assessments, including weight, blood pressure, pulse and adverse events | Every eight weeks, up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Kohut, DMD, Study Director — Pfizer
Locations (15):
- United States (15):
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Vallejo, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Fridley, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah